CLINICAL TRIAL: NCT04101851
Title: Omission of Sentinel Lymph Node Biopsy in Triple-negative and HER2-positive Breast Cancer Patients with Radiologic and Pathologic Complete Response in the Breast After Neoadjuvant Systemic Therapy: a Single-arm, Prospective Surgical Trial.
Brief Title: Omission of SLNB in Triple-negative and HER2-positive Breast Cancer Patients with RCR and PCR in the Breast After NAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toralf Reimer, MD PhD (Other)
Collaborators: European Breast Cancer Research Association of Surgical Trialists (Network); University Medicine Rostock, Rostock, Germany (sponsor) (Unknown); Else Kröner-Fresenius-Stiftung (funding) (Unknown); German Society of Senology (funding) (Unknown)
Responsible Party: Sponsor-Investigator, Toralf Reimer, MD PhD, Deputy director, Department of Obstetrics and Gynecology, University of Rostock
Organization: University of Rostock (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUBREAST-01
Record Dates: First submitted 2019-09-21; First posted 2019-09-24 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Female; Breast Cancer
Keywords: sentinel lymph node biopsy; neoadjuvant systemic therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- No axillary SLNB (Experimental): After radiologic complete remission at the end of NAST all patients will be treated with breast-conserving surgery alone without any axillary surgery. Approximately 80% of these patients will be assigned to the single study arm (no axillary SLNB) due to breast pCR (ypT0/ypTis) at the final pathology of lumpectomy.
  Interventions: Procedure: omission of SLNB

INTERVENTIONS:
Procedure: omission of SLNB — After radiologic complete remission at the end of NAST all patients will be treated with breast-conserving surgery alone without any axillary surgery.

SUMMARY:
Currently, axillary surgery for breast cancer is considered as staging procedure that does not seem to influence breast cancer mortality, since the risk of developing metastasis depends mainly on the biological behaviour of the primary (seed-and-soil model). Based on this, the postsurgical therapy should be considered on the basis of biologic tumor characteristics rather than nodal involvement.

Improvements in systemic treatments for breast cancer have increased the rates of pathologic complete response (pCR) in patients receiving neoadjuvant systemic therapy (NAST), offering the opportunity to decrease, and perhaps eliminate, surgery in patients who have a pCR.

The investigators designed a clinical trial in which only patients with the highest likelihood of having a pCR after NAST (triple-negative or HER2-positive breast cancer) will be included and type of surgery will be defined according to the response to NAST rather than on the classical T and N status at presentation. In the planned trial, axillary surgery will be eliminated completely (no axillary sentinel lymph node biopsy [SLNB]) for initially cN0 patients with radiologic complete remission (rCR) and a breast pCR as determined in the lumpectomy specimen.

The trial design is a multicenter single-arm study with a limited number of patients (N=350) which might give practice-changing results in a short period of time, sparing the time and the costs of a randomized comparison. Patients will be recruited in European countries (Austria, Germany, Italy, and Spain) over a period of 48 months.

DETAILED DESCRIPTION:
EUBREAST-01 is a prospective non-randomized, single-arm surgical trial. Included patients will be recruited for the experimental arm (no axillary SLNB in cases with breast pCR after NAST) exclusively. EUBREAST-01 is an international multicentric trial and designed by European Breast Cancer Research Association of Surgical Trialists (EUBREAST). The University Medicine Rostock (Germany) will overtake the sponsorship for the trial.

Duration of recruitment is 4 years among 36 German, 10-15 Italian, 3 Spanish, and 1 Austrian study centres. The total number of patients to be recruited into the trial will be 350. All participating centres are experienced in conduction of clinical trials and stated at least a rate of 50 primary breast cancer diagnosis per year. At least 30% of all primary breast cancer are TNBC or HER2-positive tumors. The great majority of these cases will be diagnosed in tumor stage T1-T3. The NAST with chemotherapy (plus anti-HER2 therapy if HER2-positive) is standard for this cohort in Germany, Austria, Italy, and Spain.

Efficacy analyses will be conducted after a follow-up of at least 3 years for each patient regarding the primary and for the secondary outcomes. No interim analysis is planned. Patients will be assessed for disease recurrence according to standard national clinical practice. Longest follow-up is 7 years. History and physical examination will be performed every 6 months for the first 36 months and yearly thereafter. Annual mammography and sonography will be required; other testing will be based on symptoms and investigator preference.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to breast-conserving surgery, including expected cooperation of the patients for follow-up, must be obtained and documented according to the European regulatory requirements
* Histologically confirmed unilateral primary invasive carcinoma of the breast (core biopsy). Multifocal or multicentric tumors are allowed if breast-conserving surgery is planned.
* Age at diagnosis at least 18 years
* imaging techniques with estimated tumor stage between cT1-T3 prior to NAST
* triple-negative or HER2-positive invasive breast cancer
* clinically and sonographically tumor-free axilla prior to core biopsy (cN0/iN0)
* in cases with cN0 and iN+, a negative core biopsy or fine needle aspiration (FNA) biopsy of the sonographically suspected lymph node is required
* no evidence for distant metastasis (M0)
* standard NAST with radiologic complete response (rCR)
* planned breast-conserving surgery with postoperative external whole-breast irradiation (conventional fractionation or hypofractionation)

Exclusion Criteria:

* History of malignancy within last 5 years, except curatively treated basalioma of the skin and carcinoma in situ of the cervix
* Time since last cycle of NAST >3 months (optimal <1 month)
* histologically non-invasive breast carcinoma before NAST
* ER-positive (>=10% positive cells on IHC)/HER2-negative disease (triple-positive tumors are allowed)
* cT4 or iT4 tumors
* pregnant or lactating patients
* no radiologic complete response at the end of NAST
* planned total mastectomy after NAST
* planned intraoperative radiotherapy (e.g. Intrabeam) or postoperative partial breast irradiation (e.g. multicatheter technique) alone; both procedures are allowed as boost techniques
* male patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
axillary recurrence-free survival (ARFS) after breast-conserving surgery | 3-year

SECONDARY OUTCOMES:
invasive disease-free survival | 5-year
overall survival | 5-year
locoregional disease-free survival | 5-year
  no tumor in the ipsilateral breast or ipsilateral supraclavicular, infraclavicular, internal mammary or axillary nodes
distant disease-free survival | 5-year
axillary recurrence-free survival | 5-year
Diagnostic accuracy of imaging methods for pathologic complete response (breast pCR) after NAST | 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Oreste D Gentilini, MD, Study Chair — Breast Unit, San Raffaele University and Research Hospital, Milan, Italy; Toralf Reimer, Prof., Study Chair — Department of Obstetrics and Gynecology, University of Rostock, Germany
Locations (40):
- Med. Universität Graz, Frauenklinik, Graz, Austria
- Germany (37):
  - Praxis Dres. Heinrich & Bangerter, Augsburg
  - Universitäts-Klinikum, Frauenklinik, Augsburg
  - Klinikum Mittelbaden Brustzentrum, Baden-Baden
  - DRK Kliniken Köpenick, Brustzentrum, Berlin
  - Evang. Waldkrankenhaus Spandau, Brustzentrum, Berlin
  - Sana Klinikum Lichtenberg, Berlin
  - Augusta-Klinik Brustzentrum, Bochum
  - Brustzentrum Nordsachsen, Frauenklinik, Borna
  - Marienhospital, Klinik für Gynäkologie, Bottrop
  - Kreiskliniken Böblingen, Frauenklinik, Böblingen
  - Carl-Thiem-Klinikum, Frauenklinik, Cottbus
  - Diakonissen-Krankenhaus Brustzentrum, Dresden
  - Brustzentrum Kreisklinik Ebersberg, Ebersberg
  - Uni-Klinikum Essen, Frauenklinik, Essen
  - Klinikum Esslingen, Frauenklinik, Esslingen am Neckar
  - Agaplesion Diakonie Klinikum, Frauenklinik, Hamburg
  - Albertinen Krankenhaus, Gynäkologie, Hamburg
  - Sana Klinikum Hameln-Pyrmont, Hamelin
  - Klinikum Hanau GmbH, Frauenklinik, Hanau
  - Brustzentrum Klinikum Siloah, Hanover
  - Medizinische Hochschule Hannover, Frauenklinik, Hanover
  - Universitätsklinikum Heidelberg, Frauenklinik, Heidelberg
  - ViDia Christliche Kliniken, Frauenklinik, Karlsruhe
  - Elisabeth Krankenhaus, Brustzentrum, Kassel
  - Universitäts-Klinikum Magdeburg, Frauenklinik, Magdeburg
  - Ludmillenstift, Brustzentrum, Meppen
  - Klinikum Passau, Frauenklinik, Passau
  - Universitäts-Frauenklinik am Klinikum Südstadt, Rostock
  - Helios Klinik, Gynäkologie, Schkeuditz
  - Helios Kliniken Schwerin, Frauenklinik, Schwerin
  - Diakonissen-Stiftungs-Krankenhaus, Gynäkologie, Speyer
  - Johanniter-Krankenhaus, Frauenklinik, Stendal
  - Asklepios Paulinen Klinik, Frauenklinik, Wiesbaden
  - Helios HSK, Brustzentrum, Wiesbaden
  - St. Josefs-Hospital, Frauenklinik, Wiesbaden
  - Rems-Murr-Klinik, Frauenklinik, Winnenden
  - Stadtkrankenhaus Worms gGmbH, Brustzentrum, Worms
- San Raffaele Hospital, Breast Unit, Milan, Italy
- Universidad de Navarra, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reimer T, Glass A, Botteri E, Loibl S, D Gentilini O. Avoiding Axillary Sentinel Lymph Node Biopsy after Neoadjuvant Systemic Therapy in Breast Cancer: Rationale for the Prospective, Multicentric EUBREAST-01 Trial. Cancers (Basel). 2020 Dec 9;12(12):3698. doi: 10.3390/cancers12123698. PMID 33317077
- See also: Related Info — https://eubreast.com